CLINICAL TRIAL: NCT05554588
Title: A Randomized Trial of Intrathrombus Thrombolysis Versus Aspiration Thrombectomy During Primary Percutaneous Coronary Intervention in ST-segment Elevation Myocardial Infarction Patients With High Thrombus Burden
Brief Title: Intrathrombus Thrombolysis Versus Aspiration Thrombectomy During Primary PCI
Acronym: ATTRACTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingang Zheng, Director of Cardiology, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSCF2021B02
Record Dates: First submitted 2022-09-08; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Percutaneous Coronary Intervention
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathrombus thrombolysis (Active Comparator): Intrathrombus thrombolysis with microcatheter or pierced bolloon during PPCI
  Interventions: Procedure: Intrathrombus Thrombolysis During Primary PCI
- Aspiration thrombectomy (Active Comparator): Aspiration thrombectomy during PPCI
  Interventions: Procedure: Aspiration Thrombectomy During Primary PCI

INTERVENTIONS:
Procedure: Intrathrombus Thrombolysis During Primary PCI — Intrathrombus Thrombolysis During Primary PCI
  Arms: Intrathrombus thrombolysis
Procedure: Aspiration Thrombectomy During Primary PCI — Aspiration Thrombectomy During Primary PCI
  Arms: Aspiration thrombectomy

SUMMARY:
This is an multicenter, randomized, controlled, parallel group study. ST-Segment Elevation Myocardial Infarction (STEMI) patients with high thrombus burden(HTB) will be allocated to one of the following: intrathrombus thrombolysis or manual aspiration thrombectomy during primary percutaneous coronary intervention(PPCI).

DETAILED DESCRIPTION:
The hypothesis for ATTRACTIVE trial is that the intrathrombus thrombolysis with microcatheter or pierced balloon compared to manual aspiration thrombectomy will reduce the incidence of major adverse cardiovascular events(MACEs), including cardiovascular death, recurrent myocardial infarction, cardiogenic shock, or heart failure rehospitalization, stent thrombosis and target-vessel revascularization at 1 year in STEMI patients with HTB undergoing PPCI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with:

   * Symptoms of myocardial ischemia lasting for ≥ 30 minutes AND
   * Definite ECG changes indicating STEMI: ST elevation of greater than 0.1 mV in two contiguous limb leads or 0.2 mV in two contiguous precordial leads
2. Referred for PPCI
3. Within 12 hours of symptom onset, or 12-24 hours but still suffered from persistent symptom, hemodynamic instability or fatal arrhythmia
4. High thrombus burden:

   * TIMI thrombus grade 3 or 4 after emergency coronary angiography
   * Or TIMI thrombus grade ≥3 after guidewire crossing or 1.5mm-diameter predilating the culprit lesion if emergency coronary angiography shows TIMI thrombus grade 5
5. Informed consent

Exclusion Criteria:

1. Rescue PCI after systemic thrombolysis
2. Previous CABG history
3. Life expectancy<1 year
4. Active bleeding in past 6 months, hemorrhagic disorders and prone to bleeding
5. Serious hepatic or kidney dysfunction
6. Pregnancy and lactation
7. Uncontrolled hypertension (>180/100mmHg)
8. Previous hemorrhagic stroke or ischemic stroke in past 3 months
9. Cardiogenic shock or cardio-pulmonary resuscitation
10. Informed consent cannot be obtained or follow-up cannot be completed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of major adverse cardiovascular events (MACEs) | up to 180 days
  Rate of composite of cardiovascular death, recurrent myocardial infarction, cardiogenic shock, or heart failure readmission, stent thrombosis and target-vessel revascularization

SECONDARY OUTCOMES:
Rate of ischemic stroke and transient ischemic attack (TIA) | up to 30 days
  Rate of ischemic stroke and transient ischemic attack (TIA) at 30 days
Rate of major bleeding evens (BARC type 2, 3 and 5) | up to 30 days
  Rate of major bleeding evens (BARC type 2, 3 and 5) at 30 days
Rate of key net benefit outcome | up to 1 year
  cardiovascular death, recurrent myocardial infarction, cardiogenic shock, or heart failure readmission, stent thrombosis, target-vessel revascularization, stroke and major bleeding evens (BARC 2,3 and 5)

OTHER OUTCOMES:
Rate of primary outcome at 30 days and 1 year | up to 1 year
  Rate of composite of cardiovascular death, recurrent myocardial infarction, cardiogenic shock, or heart failure readmission, stent thrombosis and target-vessel revascularization at 30 days and 1 year
Rate of individual components of primary outcome | up to 1 year
  Rate of cardiovascular death, recurrent myocardial infarction, cardiogenic shock, or heart failure readmission, stent thrombosis and target-vessel revascularization assessed separately at 30 days, 180 days and 1 year
Rate of all-cause mortality | up to 1 year
  Rate of all-cause mortality
Percentage of myocardial blush grade(MBG) of 0 or 1 | up to 30 days
  Percentage of MBG 0 or 1
Percentage of ST-segment resolution above 70% | up to 30 days
  Percentage of ST-segment resolution above 70%
Percentage of TIMI flow grade 3 | up to 30 days
  Percentage of TIMI flow grade 3
Incidence of side branch occlusion | up to 30 days
  Incidence of side branch occlusion
Incidence of distal embolism | up to 30 days
  Incidence of distal embolism
Rate of target vessel dissection | up to 30 days
  Rate of target vessel dissection assessed by coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Jingang Zheng, Doctor, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Z, Sheng Z, Che W, An S, Sun D, Zhai Z, Zhao X, Yang Y, Meng Z, Ye Z, Xie E, Li P, Yu C, Gao Y, Xiao Z, Wu Y, Dong F, Ren J, Zheng J. Design and rationale of the ATTRACTIVE trial: a randomised trial of intrAThrombus Thrombolysis versus aspiRAtion thrombeCTomy during prImary percutaneous coronary interVEntion in ST-segment elevation myocardial infarction patients with high thrombus burden. BMJ Open. 2023 Nov 10;13(11):e076476. doi: 10.1136/bmjopen-2023-076476. PMID 37949622